CLINICAL TRIAL: NCT05432258
Title: Evaluation of the Nano-Hybrid and Bulk-Fill Resin Composites: Randomised Controlled Clinical Study
Brief Title: Nano-Hybrid vs Bulk-Fill Resin Composites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Funda Cagırır Dindaroglu, Asst. Prof., Izmir Katip Celebi University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E.728477
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Composite Resin; Dental Caries in Children

STUDY DESIGN:
Intervention Model Description: In a split-mouth design, 89 patients' 2 mandibular first molars were divided into 2 groups. Per patient, one mandibular first molar had bulk-fill ormocer-based composite resin restoration and 1 mandibular first molar had nanofill composite resin restoration via incremental technic.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bulk-fill composite resin (Experimental): Bulk-fill Ormocer composite resin restorations on the mandibular first molars applied in layers of 4 mm depth
  Interventions: Device: Bulk-fill composite resin
- Nano-fill composite resin (Active Comparator): Nano-fill composite resin restorations on the mandibular first molars were applied in layers of 2 mm depth
  Interventions: Device: Nano-fill composite resin

INTERVENTIONS:
Device: Bulk-fill composite resin — Restoration of the mandibular first molars with bulk-fill composite resin as the manufacturer advises after the cavity preparation
  Other Names: Admira Fusion x-tra (Voco GmbH, Cuxhaven, Germany)
  Arms: Bulk-fill composite resin
Device: Nano-fill composite resin — Restoration of the mandibular first molars with nano-fill composite resin as the manufacturer advises after the cavity preparation
  Other Names: Grandio (Voco , Cuxhaven, Germany)
  Arms: Nano-fill composite resin

SUMMARY:
The aim of this study is to compare the 2-year clinical performance of bulk-fill composites, which can be applied as a single layer, and the nano-hybrid filled composite resins, which are frequently used in clinical routine, in children in a split-mouth design.

This study was conducted on 89 patients aged 6-12 years who had caries on bilateral mandibular first molars. Our study has a randomized, cross-controlled, and double-blind design. In split-mouth design, restorations of mandibular permanent molars completed with nano-hybrid ORMOCER based bulk-fill filling material Admira Fusion x-tra (Voco GmbH, Cuxhaven, Germany) and nano-hybrid composite Grandio (Voco , Cuxhaven, Germany). Futurabond U single dose (Voco, Cuxhaven, Germany) universal adhesive was used for all restorations, in the selective enamel etching mode. The clinical success of the restorations will be evaluated at 6, 12 and 24-month controls. Evaluations has been made by two physicians other than the one who did the restoration, who do not know which restorative material was applied to which tooth.

ELIGIBILITY:
Inclusion Criteria:

* Black class I or II caries on two bilateral mandibular permanent molars; clinically at score 3, 4 and 5 according to the ICDAS II (International Caries Detection and Evaluation System); and radiographically; with D2-RB4 and D3-RC5 levels
* plaque index (Silnes and Löe, 1964) scores of the teeth to be processed was 0 and 1
* the gingival index (Löe and Silness, 1963) score was 0

Exclusion Criteria:

* On the teeth to be processed; color change in the pits and fissures of the tooth, with no signs of caries after air drying for 5 seconds (ICDAS II Scale score 0), discoloration or opacity that is not visible when moist but observed after drying (ICDAS II Scale score 1), observable when both moist and dry or with opacity (ICDAS II Scale score 2), containing more than half of the tooth, with a large cavity in which dentin is observed (ICDAS II Score 6), Black class I and/or class II enamel-dentin caries,
* The values accepted in the evaluation of radiographic dental caries in the teeth for which the procedure is planned are E0-R0 (no radiolucency), E1-RA1 (radiolucency in the upper ½ of the enamel), E2-RA2 (radiolucency extending to the radiolucency-enamel-dentin junction in the lower ½ of the enamel) , with D1-RA3 (radiolucency observed in the upper 1/3 of the dentin),
* Non-antagonist of the teeth to be processed,
* In the gingival region of the teeth to be treated, there are areas covered with plaque from thin to medium thickness (plaque index score 2) and areas where the plaque thickness fills the gingival sulcus and where the soft attachment is high (plaque index score 3) (Löe and Silness, 1964),
* Bleeding and inflammation in the gingiva of the tooth to be treated (gingival index score (Löe and Silness, 1963) 1,2 and 3),
* Devitalized teeth for which the procedure is planned,
* The patient's lack of cooperation and physician cooperation to have the procedures performed (Score 1 and 2 on the Frankl behavioral scale).
* Having any systemic disease that prevents the treatment (ASA 2,3,4,5,6)
* Patients who will not comply with their appointments will not be included in the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Comparison of clinical performances between two restorative materials according to World Dental Federation (FDI)(1-5 scale; 1 best, 5 worst) | immediately after restoration and 24 months control
  Change of World Dental Federation (FDI) scores of restoration from baseline to 2 year
Comparison of clinical performances between two restorative materials according to US Public Health Service (USPHS) criteria (Alfa-best, Bravo, Charlie-worst) | immediately after restoration and 24 months control
  Change of the US Public Health Service (USPHS) scores of restoration from baseline to 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)